#### The GlaxoSmithKline group of companies

| Division | Worldwide Development |
|------------------|-----------------------------------|
| Information Type | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for A Randomized, Open-label, Active-Controlled, Parallel-Group, Exploratory Study on the Effects of Repeated Doses of Albiglutide compared to Exenatide on Gastric Myoelectrical Activity and Gastric Emptying in Subjects with Type 2 Diabetes Mellitus |
|---|---|---|
| <b>Compound Number</b> | : | GSK716155 |
| Effective Date | : | 17-Aug-2017 |
| Amendment | : | 01 |

### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 204879.
- This RAP is intended to describe the exploratory endpoints for the study Part A only.
- This study is terminated early prior to completion of Part A with a limited number of subjects (N=4) enrolled. Therefore, a synoptic CSR is planned and a brief RAP document is prepared accordingly.
- This RAP will be provided to the study team members to convey the content of the final Statistical Analysis Complete (SAC) Deliverable.

#### The GlaxoSmithKline group of companies

#### **Revision Chronology**

| GlaxoSmithKline<br>Document | Date | Version |
|---|---|---|
| Reporting and Analysis Plan (RAP)204879_Final | 23-Jun-2017 | Original |
| Reporting and Analysis Plan (RAP)204879_Amendment_Final_01 | 17-Aug-2017 | Amendment No. 1 |

Changes reflected in RAP Amendment No. 1 have been included to address the following:

- Appendix 5 Section 9.5.1 Data Display Numbering is updated with the appropriate listing number.
- Appendix 5 Section 9.53 added 5 listing below:
  - Listing 15: Listing of Exposure Data
  - Listing 17: Listing of Visual Analogue Scale (VAS) Scores (0-100mm scale)
  - Listing 18: Listing of Gastric Emptying 13C Excreted in Breath (kPCD1) Over Time by Treatment and Visit
  - Listing 19: Listing of Time to Half Gastric Emptying (GET1/2) by Visit
  - Listing 20: Listing of Volume of Water Ingested during EGG with Water Load Test

And Listing of all EGG Endpoints the listing number changed from 15 to 16

#### **Author's Name and Functional Area:**

| PPD | | 17 Aug 2017 |
|-----------------------|---|-------------|
| Principle Statisticia | 1 | 17-Aug-2017 |

#### Approved electronically via email by:

| PF | PPD | 17 Aug 2017 |
|----|------------------------------|-------------|
| D | Dir Statistics & Programming | 17-Aug-2017 |

### **TABLE OF CONTENTS**

| | | P | AGE |
|---|---|---|---|
| 1. | REPO | ORTING & ANALYSIS PLAN SYNPOSIS | 5 |
| 2. | CLIMA | MARY OF KEY PROTOCOL INFORMATION | 7 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | | |
| | 2.2. | Study Objective(s) and Endpoint(s) Study Design | |
| | 2.5. | 2.3.1. Overview of Study Design and Key Features | a |
| | | 2.3.2. Study Design | 9<br>0 |
| | | 2.5.2. Study Design | 9 |
| 3. | PLAN | NED ANALYSES | 10 |
| | 3.1. | Interim Analyses | 10 |
| | 3.2. | Final Analyses | 10 |
| 4. | ANAL | YSIS POPULATIONS | 10 |
| 5. | CONS | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CON\ | /ENTIONS | |
| | 5.1. | Reporting Conventions | 11 |
| 6. | STUD | DY POPULATION ANALYSES | 13 |
| 0. | 6.1. | Overview of Planned Analyses | |
| | 6.2. | Demographic and Baseline Characteristics | |
| | 6.3. | Exposure to Study Drug | |
| | 6.4. | Medications | |
| | 6.5. | Safety Analyses | |
| | 0.0. | 6.5.1. Overview of Planned Analyses | |
| | | 6.5.2. Adverse Events | |
| | | 6.5.3. Clinical Laboratory Evaluations | |
| | | 6.5.3.1. Chemistry, Hematology and Urinalysis | |
| | | 6.5.4. Vital Signs | |
| | | 6.5.5. Gastroparesis Cardinal Symptom Index Daily Dairy | |
| | | (GCSI-DD) | 16 |
| 7. | OTUE | ER STATISTICAL ANALYSES (EXPLORATORY) | 17 |
| Ι. | 7.1. | Overview of Planned Analyses | |
| | 7.1.<br>7.2. | Exploratory Analyses | |
| 8. | RFFF | RENCES | |
| 9. | | NDICES | |
| | 9.1. | Appendix 1: Time & Events | |
| | 0.0 | 9.1.1. Protocol Defined Time & Events Part A | |
| | 9.2. | Appendix 2: Assessment Windows | |
| | 0.0 | 9.2.1. Definitions of Study Day | |
| | 9.3. | Appendix 3: Values of Potential Clinical Importance | |
| | 0.4 | 9.3.1. Laboratory | |
| | 9.4.<br>0.5 | • • | |
| | 9.5. | Appendix 5: List of Data Displays 9.5.1. Data Display Numbering | |
| | | a.s. i. Data Display Nullibelling | 20 |

| 9.5.2. | Study Population Tables | 28 |
|--------|-------------------------|----|
| | Listings | |

## 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Purpose | To gain insight into a potential peripheral mechanism of nausea associated with glucagon-like peptide-1 receptor (GLP-1R) agonists; this study will compare the effect of albiglutide and exenatide on gastric myoelectrical activity (GMA), gastric emptying (GE) and nausea [as measured by visual analogue scale (VAS)] in subjects with type 2 diabetes mellitus (T2DM). The study is divided in two parts. Part A will characterize the GMA, GE and nausea response to exenatide and confirm exenatide as a positive control for Part B. At the time the RAP preparation, the study had terminated early with a limited number of subjects enrolled in Part A. |
|---|---|
| Protocol | This RAP is based on the protocol amendment 1 [(Dated: 23/June/2016) of study GSK 204879 (GSK Document No. : 2015N255772_01) and eCRF Version 1. |
| Primary<br>Objective | To evaluate the effect of exenatide on GMA (pilot phase). |
| Primary<br>Endpoint | <ul> <li>(All endpoints for Part A are exploratory)</li> <li>Change from baseline of electrogastrogram (EGG) parameters at each recording time interval (pre-and 10, 20 and 30 min after water load) compared to baseline:</li> <li>Distribution of average power by frequency region (as % of power)</li> <li>Ratios of average power post- WLT/pre-WLT by frequency region</li> <li>Percentage (%) of time with the dominant EGG frequencies in the four frequency ranges (bradygastria, normal, tachygastria and duodenal)</li> <li>Change from baseline EGG parameters related to VAS of nausea at each recording time interval (pre-and 10, 20 and 30 min after water load) at Day 4</li> </ul> |
| Study<br>Design | <ul> <li>This is a single arm, open label pilot phase to evaluate the effect of 5-day repeated doses of exenatide (10 μg twice daily) on GMA, GE and nausea in subjects with T2DM.</li> <li>The study will comprise 3 study periods: screening/wash-out (up to 3 weeks), treatment (5 days), and post-treatment follow-up (within 7 days after the last dose of exenatide).</li> <li>The study will recruit subjects with T2DM (&gt;6 months since diagnosis) with glycated hemoglobin (HbA1c) &gt;6.5% and ≤9.0%, fasting plasma glucose (FPG) &lt;=210 mg/dL (central lab) at screening and on a current regimen of diet and exercise or a stable dose of one oral anti-diabetic medication (OAM) (maintained for &gt;= 2 months prior to screening).</li> <li>Fasting capillary blood glucose will be confirmed to be &lt;=230 mg/dL at baseline.</li> <li>Subjects receiving monotherapy with an OAM of metformin,</li> </ul> |

| | <ul> <li>sulfonylurea, sodium glucose co-transporter-2 (SGLT2) inhibitors, or meglitinide at screening will be washed out for 2 days for immediate release and 4 days for extended release OAM prior to baseline.</li> <li>Subject's nutritional plan will be optimized prior to baseline and maintained during the entire study.</li> <li>All evaluations and assessments will be performed as outpatient visits. Subjects will undergo 2 EGG and 2 gastric emptying breath tests (GEBT) assessments.</li> <li>At the end of the Part A, subjects previously on an OAM will restart OAM at the discretion of the investigator after the last dose of exenatide. The half-life of exenatide (2-3 hours) should be taken into consideration.</li> <li>The total duration of a subject's participation will be approximately 5 weeks.</li> </ul> |
|---|---|
| Planned<br>Analyses | • Part A: Final Analysis: After at least 10 evaluable subjects defined as having at least one valid pre-dose EGG and one valid post –dose EGG, the final analysis for the clinical study report will be performed. At this time, the database will be frozen. The study is terminated early with a limited number of subjects enrolled in Part A. |
| Analysis<br>Populations | The analysis set will include subjects who have taken at least one dose of study medication and one valid EGG data. Data will be assessed and reviewed by the central reader before it is considered valid. |
| Hypothesis | No formal statistical hypotheses are being tested in Part A. Part A will be a pilot phase investigating the effect of repeated doses of exenatide on GMA, GE, and VAS of nausea. |
| Primary<br>Analyses | No formal statistical analyses will be performed for the exploratory endpoints for Part A. All exploratory endpoints will be assessed using descriptive statistics and graphical displays as appropriate. |

### 2. SUMMARY OF KEY PROTOCOL INFORMATION

### 2.1. Changes to the Protocol Defined Statistical Analysis Plan

The study terminated early with a limited number of subjects enrolled in Part A. Therefore, only data listings will be produced for selected data. These are limited in scope compared to the originally planned statistical analysis specified in the protocol amendment 1 [(Dated: June 23, 2016)].

### 2.2. Study Objective(s) and Endpoint(s)

#### Part A:

| Objectives | Endpoints |
|---|---|
| Exploratory Objectives | Exploratory Endpoints |
| To assess the effect of exenatide on To assess the effect of exenatide on | <ul> <li>Change from baseline of EGG parameters at each recording time interval (pre-and 10, 20 and 30 min after water load) compared to baseline:</li> <li>Distribution of average power by frequency region (as % of power)</li> <li>Ratios of average power post-WLT/pre-WLT by frequency region</li> <li>Percentage (%) of time with the dominant EGG frequencies in the four frequency ranges (bradygastria, normal, tachygastria and duodenal)</li> <li>Change from baseline EGG parameters related to VAS of nausea at each recording time interval (pre-and 10, 20 and 30 min after water load) at Day 4</li> <li>Change from baseline of time to half gastric</li> </ul> |
| GE | <ul> <li>emptying (GEt½) at Day 5</li> <li>Change from baseline of profiles of 13C excreted in breath (kPCD1) at Day 5 and at each time interval (45, 90, 120, 150, 180 and 240 min).</li> </ul> |
| To assess the volume of water | Change from baseline of volume of water ingested |
| ingested during EGG To evaluate the effect of exenatide on stomach fullness, hunger, bloating and abdominal pain during EGG with water load test To evaluate safety and tolerability of exenatide | during EGG with water load test at Day 4. Change from baseline of VAS of stomach fullness, hunger, bloating and abdominal pain during the EGG water load test at each time interval (pre-and 10, 20 and 30 min after water load) at Day 4 • Vital signs, clinical laboratory tests, AEs, and GCSI-DD. • Nausea AEs presenting outside the timing of the WLT and GCSI-DD. |

| Objectives | Endpoints |
|---|---|
| To evaluate change in gastric | At Day 4; over 30 min and at each |
| rhythm status (Data | time interval (pre-and 10, 20 and 30 min after |
| permitting) | • water load). |
| | <ul> <li>Number and % of subjects with a shift in gastric rhythm status.</li> <li>Number and % of subjects by gastric rhythm status at each time interval.</li> <li>Mean and mean change from baseline in</li> </ul> |
| | average dominant frequency |

<sup>&</sup>lt;sup>1</sup> Percent dose excreted of <sup>13</sup>C \*1000

### 2.3. Study Design

### 2.3.1. Overview of Study Design and Key Features



Due to early termination the entirety of the study conduct was not carried out.

### 2.3.2. Study Design

Part A is a single arm, open label pilot phase to evaluate the effect of 5-day repeated doses of exenatide (10 µg twice daily) on GMA, GE and nausea in subjects with T2DM. Part A will comprise 3 study periods screening/wash-out (up to 3 weeks), treatment (5±1 days), and post-treatment follow-up (within 7 days after the last dose of exenatide).

At the time the RAP is being prepared, the study is terminated early with a limited number of subjects enrolled in Part A.

### 3. PLANNED ANALYSES

### 3.1. Interim Analyses

No interim analysis is planned for this study.

### 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential step:

1. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

### 4. ANALYSIS POPULATIONS

| Part A: | Comprise of all subjects who have taken | Pharmacodynamic |
|---|---|---|
| Pharmacodynami | at least one dose of study medication and | |
| c | one valid EGG data Data will be assessed | |
| | and reviewed by the central reader before | |
| | it is considered valid. The central reader | |
| | will provide the valid data that will be | |
| | used for the analyses. | |
| All Subjects | All subjects with at least one dose of | Safety |
| | study medication. | |
| Enrolled | All enrolled subjects. | Enrolled |

#### NOTES:

 Please refer to Appendix 5: List of Data Displays which details the population to be used for each displays being generated.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

### 5.1. Reporting Conventions

- All data displays will be presented according to the Integrated Data Standards Library (IDSL) reporting standards, where applicable.
- Analyses will be performed using the 9.1.3 version of the SAS System or higher (SAS is a registered trademark of the SAS Institute Inc., Cary, NC, USA). Programs will be imported into HARP and the final output will be produced by running drivers in HARP.
- Data collected at unplanned (i.e. unscheduled) time points will not be included in the summaries by visit unless otherwise stated. Unscheduled or unplanned readings will be presented in the listings and they will be included when determining worst-case flagging for post-baseline summaries.
- In all data displays, planned and actual relative times will be relative to the study drug dosing time of the relevant dosing session.
- Refer to IDSL standards (when applicable) for decimal place conventions. Raw data will generally be presented to the same number of decimal places as it was collected.
- All data will be reported according to the actual treatment the subject received.
   Any departures from the planned treatment according to the randomization schedule will be documented in the report.
- All observations that occurred prior to dosing will be considered as part of the pre-dose period. All observations that occur during dosing will be attributed to the subject's treatment.

Deviations from the analyses in the RAP will be identified in the final clinical study report.

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

## Table 1 Overview of Appendices

| Section | Component |
|---------|-----------------------------------------------------|
| 9.1 | Appendix 1: Time & Events |
| 9.2 | Appendix 2: Assessment Windows |
| 9.3 | Appendix 3: Values of Potential Clinical Importance |
| 9.4 | Appendix 4: Abbreviations and Trademarks |
| 9.5 | Appendix 5: List of Data Displays |

#### 6. STUDY POPULATION ANALYSES

### 6.1. Overview of Planned Analyses

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 5: List of Data Displays.

Table 2 Overview of Planned Study Population Analyses

| Display Type | Data Display's Generated | | |
|---|---|---|---|
| | Figure | Table | Listing |
| Subject Disposition | | | |
| Reasons for Withdrawal from Study | | Υ | Y |
| Demography and Baseline Characteristics | | | |
| Demographics and Baseline Characteristics | | Y | Y |
| Race & Racial Combinations | | Y | Y |
| Number of subjects by Site ID | | Y | Y |
| Age Ranges | | Υ | |
| Medical Condition & Concomitant Medications | | | |
| Concomitant Medication | | | Y |
| Exposure | | | |
| Exposure to Study Drug | | | Υ |

**Note:** additional tables, listings and figures will be provided in Appendix 5: List of Data Displays.

Following review of the data, additional analyses maybe conducted to further support the evaluation and interpretation of the data.

# 6.2. Demographic and Baseline Characteristics

Continuous variables such as age, body mass index, weight, and height will be summarized using descriptive statistics (n, mean, standard deviation, and median, minimum, maximum). Categorical variables including sex, race, ethnicity, and baseline weight category (<90 kg or ≥90 kg) will be summarized using numbers and percentages. Continuous variables such as age, body mass index, weight, and height will be presented in a by-subject listing. Listings will be presented using the safety population, if appropriate.

### 6.3. Exposure to Study Drug

A by-subject listing of study drug administration will also be presented. Overall study drug administration and treatment compliance will be present with the exposure to study drug listing.

Y = Yes display generated.

### 6.4. Medications

Any prior and concomitant medication used during the study will be recorded and coded using GSKDrug Dictionary (GSKDRUG), which will be updated whenever available throughout the life of the study.

Any medication used during the study will be recorded, which will be updated whenever available throughout the life of the study.

All medications will be listed.

### 6.5. Safety Analyses

#### 6.5.1. Overview of Planned Analyses

The safety analyses will be based on all subjects' population.

Table 3 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 5: List of Data Displays.

Table 3 Overview of Planned Safety Analyses

| | | Obse | erved | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| Endpoints | Summary | | Individual | | Summary | | Individual | |
| | T | F | F | L | Т | F | F | L |
| Adverse Events | Υ | | | Υ | | | | |
| Clinical Laboratory | | | | Υ | | | | |
| Vital Signs | | | | Υ | | | | |
| GCSI-DD | | | | Υ | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

Following review of the data, additional analyses maybe conducted to further support the evaluation and interpretation of the data.

#### 6.5.2. Adverse Events

All AEs will be coded using MedDRA which will be updated whenever available throughout the life of the study.

All AEs will be listed in a subject data listing.

#### 6.5.3. Clinical Laboratory Evaluations

### 6.5.3.1. Chemistry, Hematology and Urinalysis

Laboratory parameters include the following tests: hematology, chemistry and urinalysis. Established or generally acknowledged methods, normal ranges, and quality control procedures will be supplied by central lab for the study records.

Hematology parameters include red blood count, hemoglobin, hematocrit white blood cell count with differential, and platelet count. Chemistry blood urea nitrogen (BUN), potassium, aspartate aminotransferase (AST), total and direct bilirubin, creatinine, sodium, ALT, total protein, calcium, magnesium, chloride, phosphorus albumin, gamma glutamyl transferase (GGT), estimated glomerular filtration rate (eGFR), and lipids

(including total cholesterol, LDL-C, HDL C, triglycerides,). Urinalysis parameters include microalbumin and creatnine and specific gravity, pH, glucose, nitrates, leukocytes esterase, blood and ketones by dipstick and microscopic examination (if blood or protein is abnormal).

All laboratory parameters as collected will be presented in by-subject listings at every scheduled assessment time point. All listings will be done for the safety population and all laboratory data will be listed including other laboratory tests, such as TSH, and urine pregnancy test results.

Additionally, the number of subjects with laboratory values of potential clinical concern will be provided in a listing by treatment group and scheduled assessment time point for hematology and chemistry. The criteria for laboratory values of potential clinical concern are detailed in Appendix 3: Values of Potential Clinical Importance.

A listing of laboratory values of potential clinical concern will be provided for liver function tests, including ALT, AST, and total bilirubin. The criteria for liver function tests of potential clinical concern are detailed in Appendix 3: Values of Potential Clinical Importance.

### 6.5.4. Vital Signs

The vital sign analysis will include systolic blood pressure (mmHg), diastolic blood pressure (mmHg), and heart rate (bpm).

Each vital sign parameter at every scheduled assessment time point will be presented in by-subject listings.

All listings will be produced for all subjects population.

#### 6.5.5. Gastroparesis Cardinal Symptom Index Daily Dairy (GCSI-DD)

The GCSI-DD consists of nine symptom severity items covering the following domains: nausea/vomiting; fullness/early satiety, and bloating. In addition, the GCSI-DD contains two symptom severity items upper abdominal pain and overall rating of gastroparesis symptoms. Patients rate each symptom on a 6-point scale from 0-5 with lower scores representing less symptom severity. All questions addressed in the GCSI-DD and the overall severity question will be listed in a subject data listing and by time point.

## 7. OTHER STATISTICAL ANALYSES (EXPLORATORY)

### 7.1. Overview of Planned Analyses

The study was terminated early and therefore no analysis will be performed but data listing will be generated for all exploratory endpoints as in Appendix 5.

### 7.2. Exploratory Analyses

Listing will be provided for all endpoints.

## 8. REFERENCES

None.

## 9. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 9.1 | Appendix 1: Time and Events |
| Section 9.2 | Appendix 2: Assessment Windows |
| Section 9.3 | Appendix 3: Values of Potential Clinical Importance |
| Section 9.4 | Appendix 4: Abbreviations & Trade Marks |
| Section 9.5 | Appendix 5: List of Data Displays |

#### 9.1. **Appendix 1: Time & Events**

#### 9.1.1. Protocol Defined Time & Events Part A

| Procedures | Screening/Wash-Out Period<br>(0-3 Weeks) | | | Treatment Period (exenatide)<br>(5 Days) | | | | | Un-<br>schedule | Early | Follow Up |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | -21 to<br>Day -4 | Day -3<br>to -5 | Day -113 | Day 1 | Day 2 | Day 3 | Day 4<br>± 1 day <sup>13</sup> | Day 5<br>± 1 day <sup>13</sup> | d | Withdrawal | Within 7<br>Days |
| Study Visit | 1 | | 2 | 3 | 3 | 8 8 | 4 | 5 | | | 6 |
| Informed consent | X | | | | | | | | | | |
| Inclusion and exclusion criteria | X | · · | χ1 | | ii . | | | i i | | i i | |
| Demography, medical/disease history | X | Š. | | | | | į. | | | | |
| Enrolment into Treatment Phase | | | | X | | | | | | | |
| OAM washout <sup>2</sup> | | Х | | | | | | | | | |
| GEBT <sup>3</sup> | 7 | | X | | 9 | | | X12 | | | |
| EGG /water load / VAS3 | | | | χ11 | | | X12 | | | | |
| ECG | X | | | | | | | | | | |
| Vital Signs | X | | X | X | i i | | X | X | | X | X |
| Height, Weight, BMI | X | * | | | | | | | | | |
| Physical exam (F, Full; B, Brief)4 | F | | | 6 | | 8 8 | | В | | В | |
| Concomitant medications review | X | | X | X | | | X | | X | X | Х |
| AEs, SAEs, AEs of special interest review | X5 | | χ5 | X | ĵ | | X | X | X | X | X |
| PAGI-SYM <sup>6</sup> | X | W | | ii. | 1 | | | | | * | |
| GCSI-DD | 8 | | Х | X | | | X | X | | | |
| Chemistry, hematology, urinalysis, lipids7 | X | | | | | | | X | | Х | |
| HbA1c | X | ** | | | | | | | | **** | |
| FPG | X | ** | X | X | | | X | X | X | X | X |
| Fasting capillary glucose at clinic <sup>8</sup> | | | X | X | | | X | X | | | |
| Diet/Exercise/SMBG advice/reinforcement9 | X | Х | | | | | | X | X | X | X |
| Estradiol and FSH (females only: if required) | Х | | | | | | | | | | 3000 |
| Serum/Urine pregnancy test (FRP only) | S | | U | | | | | U | | U | U |
| TSH, Amylase and lipase | X | | | | 1 | | | | | 1000 | |
| Genetics sample <sup>10</sup> | * | | | X | | | | | | | |
| RAMOS registration | | | | X | | | | | | X | Х |

| Procedures | | ng/Wash-O<br>(0-3 Weeks | | Treatment Period (exenatide)<br>(5 Days) | | | | Un- | Early | Follow Up | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | -21 to Day -3<br>Day -4 to -5 Day -1 | Day -113 | Day 1 | Day 2 | Day 3 | Day 4<br>±1 day <sup>13</sup> | Day 5<br>± 1 day <sup>(3)</sup> | schedule<br>d | Withdrawal | Within 7<br>Days | |
| Study Visit | 1 | | 2 | 3 | | | 4 | 5 | | | 6 |
| Exenatide dosing | | 1 | | X11 | X | X | X12 | X12 | | | |
| Study medication compliance | | 8 | | X | | | X | X | | | |

- Before baseline assessment (Day -1), the investigator must review all inclusion and exclusion criteria to confirm subject's eligibility. If a subject no longer meets all of the
  eligibility criteria, do not administer the study treatment and contact the Medical Monitor to discuss how to proceed (e.g., to determine if repeat testing is warranted).
   For subjects taking OAM at screening only. At a minimum, two day washout for immediate release and at minimum 4 day washout for extended release OAMs. See footnote
  - 13. For information on restarting OAM refer to Section 6.9.
- A small meal will be provided 2 hrs prior to the EGG procedure (Section 7.3.1). A meal will also be provided post-procedure for both the EGG and GEBT.
- Details of full and brief physical examinations are provided in Section 7.4.3.
- SAEs related to study participation only.
- The GCSI-DD questionnaire will be completed after the standard AE questions have been answered.
- Clinical chemistry, hematology, urinalysis and lipid assessments are described in Section 7.4.6. Lipids will be assessed at screening only.
- 8. Fasting capillary glucose will be measured prior to administration of exenatide. On GEBT (Day 5) or EGG (Day 1 and Day 4) assessment days, fasting capillary glucose will be measured prior to the GEBT or EGG procedure.
- 9. Subjects will be provided with diet and exercise guidance (see Section 7.4.8) and instructed on self monitoring blood glucose at screening (See Section 7.4.9). Subject will be instructed to bring in their glucometers at each visit for review. Diet/exercise/SMBG reinforced at subsequent visits.
- 10. Informed consent for optional genetic research should be obtained before collecting a sample.
- 11. On the morning of Day 1, subjects will receive instructions and training on exenatide self administration and will be monitored by medical staff at the clinic during administration of the first dose. The first dose of exenatide will be administered after the baseline EGG procedure and before the post-procedure meal.
- 12. On Day 4 and 5, the morning close of exenaticle will be administered at clinic 1 hr (±15 min) before the EGG or GEBT procedure.
- Every effort should be made to schedule the procedures on the nominal visit day identified. However, in order to meet scheduling needs, subjects taking QAM can schedule Day-1 up to 3 days prior to Day 1 and the OAM stopped at least the day before the GEBT. For subjects treated with diet and exercise alone Day-1 can occur within 7 days prior to Day 1. The EGG and GEBT should not be scheduled on the same day

Note: section noted in time and event table referring to the protocol.

## 9.2. Appendix 2: Assessment Windows

### 9.2.1. Definitions of Study Day

When study day is used for display or in comparisons the following algorithm will be used:

- Study day = date of assessment date of first dose + 1, if day of assessment >= first dose date
- Study day = date of assessment date of first dose, if day of assessment < first dose date

Note that the date of first dose is Day 1 and the day before the date of first dose is Day -1 (there is no Day 0).

# 9.3. Appendix 3: Values of Potential Clinical Importance

# 9.3.1. Laboratory

| | | Hematology | |
|---|---|---|---|
| Laboratory<br>Test | Units | Change from Baseline of Potential Clinical Concern | Potential Clinical Concern<br>Value |
| Basophils | GI/L | None | None |
| Eosinophils | GI/L | None | None |
| Hematocrit | 1 | >0.1 decrease | >0.05 below LLN<br>>0.04 above ULN |
| Hemoglobin | g/L | >25 g/L decrease | >20 g/L below LLN<br>>10 g/L above ULN |
| Lymphocytes | GI/L | None | <0.5 x LLN |
| Monocytes | GI/L | None | None |
| Neutrophils | GI/L | None | <1 GI/L |
| Neutrophil<br>Bands | GI/L | None | None |
| Platelets | GI/L | None | <80 GI/L<br>>500 GI/L |
| Red Blood Cell<br>Count | TI/L | None | None |
| Segmented<br>Neutrophils | GI/L | None | <0.5 x LLN |
| White Blood Cell<br>Count | GI/L | None | >1 GI/L below LLN<br>>5 GI/L above ULN |

| | Chemistry | | |
|---|---|---|---|
| Laboratory<br>Test | Units | Change from Baseline of<br>Potential Clinical Concern | Potential Clinical Concern<br>Value |
| Albumin | g/L | None | >5 g/L above ULN or below LLN |
| Alkaline<br>Phosphatase | U/L | None | >3 x ULN |
| ALT | U/L | None | >3 x ULN |
| AST | U/L | None | >3 x ULN |
| Bicarbonate<br>(Carbon Dioxide<br>Content) | mmol/L | None | <16 mmol/L<br>> 40 mmol/L |
| Blood Urea<br>Nitrogen | mmol/L | None | >2 x ULN |
| Calcitonin | pmol/L | None | >100 |
| Calcium | mmol/L | None | <1.8 mmol/L<br>>3.0 mmol/L |

| | | Chemistry | |
|---|---|---|---|
| Laboratory<br>Test | Units | Change from Baseline of<br>Potential Clinical Concern | Potential Clinical Concern<br>Value |
| Chloride | mmol/L | None | None |
| Creatinine | umol/L | None | >159 umol/L |
| Direct Bilirubin | umol/L | None | >1.35 x ULN |
| Gamma<br>Glutamyl<br>Transferase | U/L | None | >3 x ULN |
| Glucose<br>(fasting) | mmol/L | None | <3 mmol/L<br>>22 mmol/L |
| Magnesium | mmol/L | None | <1 mmol/L<br>>4 mmol/L |
| Phosphorus | mmol/L | None | >0.323 mmol/L above ULN or below LLN |
| Potassium | mmol/L | None | >0.5 mmol/L below LLN<br>>1.0 mmol/L above ULN |
| Sodium | mmol/L | None | >5 mmol/L above ULN or below LLN |
| Total Bilirubin | umol/L | None | >1.5 x ULN |
| Total Protein | g/L | None | >15 g/L above ULN or below LLN |
| Uric acid | umol/L | None | >654 umol/L |
| Free Fatty Acids | mmol/L | None | None |
| HDL Cholesterol | mmol/L | None | None |
| LDL Cholesterol | mmol/L | None | None |
| Triglycerides | mmol/L | None | > 9.04 mmol/L |
| Total<br>Cholesterol | mmol/L | None | None |

| Laboratory Test | Potential Clinical Concern Value |
|-----------------|-----------------------------------------|
| ALT | ≥ 2 x ULN |
| | ≥ 3 x ULN |
| | ≥ 5 x ULN |
| | ≥ 8 x ULN |
| | ≥ 10 x ULN |
| | ≥ 3 x ULN and Total Bilirubin ≥ 2 x ULN |
| AST | ≥ 2 x ULN |
| | ≥ 3 x ULN |
| | ≥ 5 x ULN |
| | ≥ 8 x ULN |
| | ≥ 10 x ULN |
| | ≥ 3 x ULN and Total Bilirubin ≥ 2 x ULN |
| Total Bilirubin | ≥ 1.5 x ULN |
| | ≥ 2 x ULN |
| | ≥ 3 x ULN |
| | ≥ 5 x ULN |
| | ≥ 8 x ULN |
| | ≥ 10 x ULN |

# 9.4. Appendix 4 – Abbreviations & Trade Marks

## Abbreviations

| ADA | American Diabetes Association |
|------------|--------------------------------------------------------|
| AE | adverse event |
| ALT (SGPT) | alanine aminotransferase (serum glutamic pyruvic |
| | transaminase) |
| AST (SGOT) | aspartate aminotransferase (serum glutamic oxaloacetic |
| | transaminase) |
| BMI | body mass index |
| BUN | blood urea nitrogen |
| CI | confidence interval |
| CONSORT | Consolidated Standards of Reporting Trials |
| CPK | creatine phosphokinase |
| CV | cardiovascular |
| DCC | dual chamber cartridge |
| DNA | deoxyribonucleic acid |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| eGFR | estimated glomerular filtration rate |
| EGG | electrogastrogram |
| ELISA | enzyme-linked immunosorbent assay |
| EMA | European Medicines Agency |
| FDA | US Food and Drug Administration |
| FFA | free fatty acids |
| FPG | fasting plasma glucose |
| FRP | females of reproductive potential |
| FSH | follicle stimulating hormone |
| GCP | Good Clinical Practice |
| GCSP | Global Clinical Safety and Pharmacovigilance |
| GGT | gamma glutamyl transferase |
| GI | gastrointestinal |
| GLP-1 | glucagon-like peptide-1 |
| GSK | GlaxoSmithKline |
| НА | human albumin |
| HbA1c | glycated hemoglobin |
| HBcAb | hepatitis B core antibody |
| HBsAg | hepatitis B surface antigen |
| HIV | human immunodeficiency virus |
| hCG | human chorionic gonadotrophin |
| HDL-c | high density lipoproteins |
| HRP | horseradish peroxidase |
| HRT | hormone replacement therapy |
| IB | Investigator's Brochure |
| ICH | International Conference on Harmonization |

| INR international normal range IP investigational product IRB Institutional Review Board ISRs injection site reactions ITT intent-to-treat IVRS Interactive Voice Response System LDH lactate dehydrogenase LDL-c low density lipoproteins; LMCF last mean carried forward K2EDTA di-potassium ethylenediaminetetraacetic acid MACE major adverse cardiovascular event MCH mean corpuscular hemoglobin MCV mean corpuscular volume MDRD Modification of Diet in Renal Disease MedDRA Medical Dictionary for Regulatory Activities MEN-2 multiple endocrine neoplasia type 2 MI myocardial infarction MSDS Material Safety Data Sheet MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SMPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | IEC | Independent Ethics Committee |
|---|---|---|
| IP investigational product IRB Institutional Review Board ISRs injection site reactions ITT intent-to-treat IVRS Interactive Voice Response System IDH lactate dehydrogenase LDL-e low density lipoproteins; LMCF last mean carried forward K2EDTA di-potassium ethylenediaminetetraacetic acid MACE major adverse cardiovascular event MCH mean corpuscular hemoglobin MCV mean corpuscular volume MDRD Modification of Diet in Renal Disease MedDRA Medical Dictionary for Regulatory Activities MEN-2 multiple endocrine neoplasia type 2 MI myocardial infarction MSDS Material Safety Data Sheet MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.e. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SMPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | | |
| IRB Institutional Review Board ISRs injection site reactions ITT interactive Voice Response System LDH lactate dehydrogenase LDL-c low density lipoproteins; LMCF last mean carried forward K <sub>2</sub> EDTA di-potassium ethylenediaminetetraacetic acid MACE major adverse cardiovascular event MCH mean corpuscular hemoglobin MCV mean corpuscular volume MDRD Modification of Diet in Renal Disease MedDRA Medical Dictionary for Regulatory Activities MEN-2 multiple endocrine neoplasia type 2 MI myocardial infarction MSDS Material Safety Data Sheet MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokineties PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell S.C. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | | |
| ISRs injection site reactions ITT intent-to-treat IVRS Interactive Voice Response System LDH lactate dehydrogenase LDL-c low density lipoproteins; LMCF last mean carried forward K2EDTA di-potassium ethylenediaminetetraacetic acid MACE major adverse cardiovascular event MCH mean corpuscular hemoglobin MCV mean corpuscular lemoglobin MCV mean corpuscular volume MDRD Modification of Diet in Renal Disease MedDRA Medical Dictionary for Regulatory Activities MEN-2 multiple endocrine neoplasia type 2 MI myocardial infarction MSDS Material Safety Data Sheet MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas TZDM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | | |
| ITT intent-to-treat IVRS Interactive Voice Response System LDH lactate dehydrogenase LDL-c low density lipoproteins; LMCF last mean carried forward K2EDTA di-potassium ethylenediaminetetracetic acid MACE major adverse cardiovascular event MCH mean corpuscular hemoglobin MCV mean corpuscular volume MDRD Modification of Diet in Renal Disease MedDRA Medical Dictionary for Regulatory Activities MEN-2 multiple endocrine neoplasia type 2 MI myocardial infarction MSDS Material Safety Data Sheet MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | | |
| IVRS Interactive Voice Response System LDH lactate dehydrogenase LDL-c low density lipoproteins; LMCF last mean carried forward K2EDTA di-potassium ethylenediaminetetraacetic acid MACE major adverse cardiovascular event MCH mean corpuscular hemoglobin MCV mean corpuscular volume MDRD Modification of Diet in Renal Disease MedDRA Medical Dictionary for Regulatory Activities MEN-2 multiple endocrine neoplasia type 2 MI myocardial infarction MSDS Material Safety Data Sheet MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SMPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | | • |
| LDH lactate dehydrogenase LDL-c low density lipoproteins; LMCF last mean carried forward K2EDTA di-potassium ethylenediaminetetraacetic acid MACE major adverse cardiovascular event MCH mean corpuscular hemoglobin MCV mean corpuscular volume MDRD Modification of Diet in Renal Disease MedDRA Medical Dictionary for Regulatory Activities MEN-2 multiple endocrine neoplasia type 2 MI myocardial infarction MSDS Material Safety Data Sheet MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus thyroid stimulating hormone ULN upper limit of normal range white blood cell white blood cell white blood cell white blood cell | | |
| LDL-c low density lipoproteins; LMCF last mean carried forward K2EDTA di-potassium ethylenediaminetetraacetic acid MACE major adverse cardiovascular event MCH mean corpuscular hemoglobin MCV mean corpuscular volume MDRD Modification of Diet in Renal Disease MedDRA Medical Dictionary for Regulatory Activities MEN-2 multiple endocrine neoplasia type 2 MI myocardial infarction MSDS Material Safety Data Sheet MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus thyroid stimulating hormone ULN upper limit of normal range white blood cell white blood cell white blood cell white blood cell white blood cell | | ÷ • |
| LMCF K2EDTA di-potassium ethylenediaminetetraacetic acid MACE major adverse cardiovascular event MCH mean corpuscular hemoglobin MCV mean corpuscular volume MDRD Modification of Diet in Renal Disease MedDRA Medical Dictionary for Regulatory Activities MEN-2 multiple endocrine neoplasia type 2 MI myocardial infarction MSDS Material Safety Data Sheet MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | | |
| K₂EDTA di-potassium ethylenediaminetetraacetic acid MACE major adverse cardiovascular event MCH mean corpuscular hemoglobin MCV mean corpuscular volume MDRD Modification of Diet in Renal Disease MedDRA Medical Dictionary for Regulatory Activities MEN-2 multiple endocrine neoplasia type 2 MI myocardial infarction MSDS Material Safety Data Sheet MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas | | low density lipoproteins; |
| MACE major adverse cardiovascular event MCH mean corpuscular hemoglobin MCV mean corpuscular volume MDRD Modification of Diet in Renal Disease MedDRA Medical Dictionary for Regulatory Activities MEN-2 multiple endocrine neoplasia type 2 MI myocardial infarction MSDS Material Safety Data Sheet MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | | |
| MCH mean corpuscular hemoglobin MCV mean corpuscular volume MDRD Modification of Diet in Renal Disease MedDRA Medical Dictionary for Regulatory Activities MEN-2 multiple endocrine neoplasia type 2 MI myocardial infarction MSDS Material Safety Data Sheet MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | | |
| MCV mean corpuscular volume MDRD Modification of Diet in Renal Disease MedDRA Medical Dictionary for Regulatory Activities MEN-2 multiple endocrine neoplasia type 2 MI myocardial infarction MSDS Material Safety Data Sheet MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | | |
| MDRDModification of Diet in Renal DiseaseMedDRAMedical Dictionary for Regulatory ActivitiesMEN-2multiple endocrine neoplasia type 2MImyocardial infarctionMSDSMaterial Safety Data SheetMTCmedullary thyroid cancerOC RDCOracle Clinical Remote Data CapturePACPancreatitis Adjudication CommitteePDpharmacodynamicsPKpharmacodynamicsPFper protocolPTS-DPMKPlatform Technologies and Science-Drug Metabolism and PharmacokineticsRAPReporting Analysis PlanRBCred blood cellRNAribonucleic acids.c.subcutaneousSACStatistical Analysis CompleteSAEserious adverse eventSmPCSummary of Product CharacteristicsSRMStudy Reference ManualSUsulfonylureasT2DMtype 2 diabetes mellitusTSHthyroid stimulating hormoneULNupper limit of normal rangeWBCwhite blood cell | | |
| MedDRA Medical Dictionary for Regulatory Activities MEN-2 multiple endocrine neoplasia type 2 MI myocardial infarction MSDS Material Safety Data Sheet MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC | MCV | |
| MEN-2 multiple endocrine neoplasia type 2 MI myocardial infarction MSDS Material Safety Data Sheet MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | MDRD | Modification of Diet in Renal Disease |
| MI myocardial infarction MSDS Material Safety Data Sheet MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | MedDRA | Medical Dictionary for Regulatory Activities |
| MSDS Material Safety Data Sheet MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | MEN-2 | multiple endocrine neoplasia type 2 |
| MTC medullary thyroid cancer OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | MI | myocardial infarction |
| OC RDC Oracle Clinical Remote Data Capture PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | MSDS | Material Safety Data Sheet |
| PAC Pancreatitis Adjudication Committee PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | MTC | medullary thyroid cancer |
| PD pharmacodynamics PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | OC RDC | Oracle Clinical Remote Data Capture |
| PK pharmacokinetics PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | PAC | Pancreatitis Adjudication Committee |
| PP per protocol PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | PD | pharmacodynamics |
| PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | PK | pharmacokinetics |
| PTS-DPMK Platform Technologies and Science-Drug Metabolism and Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | PP | per protocol |
| Pharmacokinetics RAP Reporting Analysis Plan RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | PTS-DPMK | |
| RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | | |
| RBC red blood cell RNA ribonucleic acid s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | RAP | Reporting Analysis Plan |
| s.c. subcutaneous SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | RBC | |
| SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | RNA | ribonucleic acid |
| SAC Statistical Analysis Complete SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | s.c. | subcutaneous |
| SAE serious adverse event SmPC Summary of Product Characteristics SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | | |
| SmPCSummary of Product CharacteristicsSRMStudy Reference ManualSUsulfonylureasT2DMtype 2 diabetes mellitusTSHthyroid stimulating hormoneULNupper limit of normal rangeWBCwhite blood cell | | |
| SRM Study Reference Manual SU sulfonylureas T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | | |
| SUsulfonylureasT2DMtype 2 diabetes mellitusTSHthyroid stimulating hormoneULNupper limit of normal rangeWBCwhite blood cell | | |
| T2DM type 2 diabetes mellitus TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | | |
| TSH thyroid stimulating hormone ULN upper limit of normal range WBC white blood cell | | |
| ULN upper limit of normal range WBC white blood cell | | |
| WBC white blood cell | | |
| WCBP women of child bearing potential | | |

## **Trademark Information**

| Trademarks of the GlaxoSmithKline |
|-----------------------------------|
| group of companies |

NONE

Trademarks not owned by the GlaxoSmithKline group of companies

MedDRA

# 9.5. Appendix 5: List of Data Displays

# 9.5.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Listings | Tables |
|-----------------------|----------|------------|
| Study Population | 1 to 5 | 1.1 to 1.5 |
| Safety | 6 to 15 | 1.6 to 1.7 |
| Exploratory Endpoints | 16 to 20 | |

### 9.5.2. Study Population Tables

| Stud | y Population | Tables | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| [Dis | position] | | | | |
| 1.1. | All<br>Subjects | ES1/ES1A | Summary of Subjects Disposition for the Subject Conclusion Record | | |
| [Den | nographics an | d Baseline Chara | acteristics] | | |
| 1.2. | All<br>Subjects | DM1 | Summary of Demographic Characteristics | | |
| 1.3. | All<br>Subjects | DM5 | Summary of Race & Racial Combinations | | |
| 1.4. | Enrolled | NS1 | Summary of Number of<br>Subjects by Country and Site<br>ID | | |
| 1.5. | Enrolled | DM11 | Summary of Age Ranges | | |
| Safe | ty Tables | | | | |
| 1.6. | All<br>Subjects | AE15 | Summary of Common (>=2%)<br>Non-serious AEs by System<br>Organ Class and Preferred<br>Term | | |
| 1.7. | All<br>Subjects | AE16 | Summary of Serious AEs by<br>System Organ Class and<br>Preferred Term | | |

# 9.5.3. Listings

| Listings | | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL /<br>TST ID /<br>Exampl<br>e Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 1. | All<br>Subjects | | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | |
| 2. | All<br>Subjects | | Listing of Reasons for Withdrawal from Study | | |
| 3. | All<br>Subjects | | Listing of Demographics and Baseline Characteristics | | |
| 4. | All<br>Subjects | | Listing of Race | | |
| 5. | All<br>Subjects | | Listing of Subjects by Site ID | | |
| 6. | All<br>Subjects | | Listing of Concomitant Medication by Generic Term | | |
| 7. | All<br>Subjects | | Listing of All Adverse Events | | |
| 8. | All<br>Subjects | | Listing of Hematology Laboratory Data | | |
| 9. | All<br>Subjects | | Listing of Chemistry Laboratory Data | | |
| 10. | All<br>Subjects | | Listing of Urinalysis Laboratory Data | | |
| 11. | All<br>Subjects | | Listing of Laboratory Data for<br>Subjects with Any Value of Potential<br>Clinical Concern | | |
| 12. | All<br>Subjects | | Listing of Liver Functions with Any Value of Potential Clinical Concern | | |
| 13. | All<br>Subjects | | Listing of Vital Signs | | |
| 14. | All<br>Subjects | | Listing of GCSI-DD | | |
| 15. | All<br>Subjects | | Listing of Exposure Data | | |
| 16. | Pharmaco<br>dynamic | | Listing of all EGG endpoints. | | |
| 17. | Pharmaco<br>dynamic | | Listing of Visual Analogue Scale (VAS) Scores (0-100mm scale) | | |

| Listings | | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL /<br>TST ID /<br>Exampl<br>e Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 18. | Pharmaco<br>dynamic | | Listing of Gastric Emptying 13C<br>Excreted in Breath (kPCD1) Over<br>Time by Treatment and Visit | | |
| 19. | Pharmaco<br>dynamic | | Listing of Time to Half Gastric<br>Emptying (GET1/2) by Visit | | |
| 20. | Pharmaco<br>dynamic | | Listing of Volume of Water Ingested during EGG with Water Load Test | | |

# CONFIDENTIAL The GlaxoSmithKline group of companies

204879

| Division | : Worldwide Development |
|------------------|-------------------------------------|
| Information Type | : Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for A Randomized, Open-label, Active-Controlled, Parallel-Group, Exploratory Study on the Effects of Repeated Doses of Albiglutide compared to Exenatide on Gastric Myoelectrical Activity and Gastric Emptying in Subjects with Type 2 Diabetes Mellitus |
|---|---|---|
| <b>Compound Number</b> | : | GSK716155 |
| <b>Effective Date</b> | : | 23-June-2017 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 204879.
- This RAP is intended to describe the exploratory endpoints for the study Part A only.
- This study is terminated early prior to completion of Part A with a limited number of subjects (N=4) enrolled. Therefore, a synoptic CSR is planned and a brief RAP document is prepared accordingly.
- This RAP will be provided to the study team members to convey the content of the final Statistical Analysis Complete (SAC) Deliverable.

#### **Author's Name and Functional Area:**

| PPD | | 23-June-2017 |
|------------------------|---|--------------|
| Principle Statistician | 1 | 23-June-2017 |

#### Approved by:

| PPD | 23-June-2017 |
|------------------------------|---------------|
| Dir Statistics & Programming | 23-Julie-2017 |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

204879

### **TABLE OF CONTENTS**

| | | | PA | GE |
|---|---|---|---|---|
| 1. | REPO | RTING & A | ANALYSIS PLAN SYNPOSIS | 4 |
| 2. | SLIMAN | /ΔDV ∩E k | (EY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | | to the Protocol Defined Statistical Analysis Plan | |
| | 2.2.<br>2.3. | | ijective(s) and Endpoint(s) | |
| | | | isign | |
| | 2.5. | 2.3.1. | Overview of Study Design and Key Features | |
| | | 2.3.1. | Study Design | ι |
| | | 2.5.2. | Study Design | 0 |
| 3. | PLAN | NED ANAL | YSES | 9 |
| | 3.1. | | | |
| | 3.2. | Final Ana | alyses | 9 |
| 4. | ΔΝΔΙ | VSIS POP | ULATIONS | a |
| ᅻ. | | | | 9 |
| 5. | | | ONS FOR DATA ANALYSES AND DATA HANDLING | ۵ |
| | 5.1. | | g Conventions | |
| | 0.1. | reporting | 9 0011 0110 | 0 |
| 6. | STUD | Y POPULA | ATION ANALYSES | . 10 |
| | 6.1. | Overview | of Planned Analyses | . 10 |
| | 6.2. | | phic and Baseline Characteristics | |
| | 6.3. | | to Study Drug | |
| | 6.4. | | ons | |
| | 6.5. | Safety Ar | nalyses | 12 |
| | | 6.5.1. | Overview of Planned Analyses | |
| | | 6.5.2.<br>6.5.3. | Adverse Events | |
| | | | Clinical Laboratory Evaluations | |
| | | | 6.5.3.1. Chemistry, Hematology and Urinalysis | |
| | | 6.5.4. | Vital Signs | 13 |
| | | 6.5.5. | Gastroparesis Cardinal Symptom Index Daily Dairy | |
| | | | (GCSI-DD) | . 13 |
| 7. | OTLIC | D CTATIC | TICAL ANALYCES (EVDLODATODY) | 42 |
| ١. | 7.1. | | TICAL ANALYSES (EXPLORATORY)<br>of Planned Analyses | |
| | 7.1.<br>7.2. | | ory Analyses | |
| | | · | | |
| 8. | REFE | RENCES | | . 14 |
| 9. | APPE | NDICES | | . 15 |
| | 9.1. | | (1 Time & Events | |
| | | 9.1.1. | Protocol Defined Time & Events Part A | . 16 |
| | 9.2. | Appendix | 2 Assessment Windows | |
| | | 9.2.1. | Definitions of Study Day | . 17 |
| | 9.3. | Appendix | 3 Values of Potential Clinical Importance | . 18 |
| | | 9.3.1. | Laboratory | |
| | 9.4. | Appendix | 4 – Abbreviations & Trade Marks | |
| | 9.5. | | c 5 List of Data Displays | |
| | | 9.5.1. | Data Display Numbering | . 24 |

## 2017N325664\_00

| | | 204879 |
|--------|-------------------------|--------|
| 9.5.2. | Study Population Tables | 24 |
| | Listings | |

204879

### 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Purpose | To gain insight into a potential peripheral mechanism of nausea associated with glucagon-like peptide-1 receptor (GLP-1R) agonists; this study will compare the effect of albiglutide and exenatide on gastric myoelectrical activity (GMA), gastric emptying (GE) and nausea [as measured by visual analogue scale (VAS)] in subjects with type 2 diabetes mellitus (T2DM). The study is divided in two parts. Part A will characterize the GMA, GE and nausea response to exenatide and confirm exenatide as a positive control for Part B. At the time the RAP preparation, the study had terminated early with a limited number of subjects enrolled in Part A. |
|---|---|
| Protocol | This RAP is based on the protocol amendment 1 [(Dated: 23/June/2016) of study GSK 204879 (GSK Document No. : 2015N255772_01) and eCRF Version 1. |
| Primary<br>Objective | To evaluate the effect of exenatide on GMA (pilot phase). |
| Primary<br>Endpoint | <ul> <li>(All endpoints for Part A are exploratory)</li> <li>Change from baseline of electrogastrogram (EGG) parameters at each recording time interval (pre-and 10, 20 and 30 min after water load) compared to baseline:</li> <li>Distribution of average power by frequency region (as % of power)</li> <li>Ratios of average power post- WLT/pre-WLT by frequency region</li> <li>Percentage (%) of time with the dominant EGG frequencies in the four frequency ranges (bradygastria, normal, tachygastria and duodenal)</li> <li>Change from baseline EGG parameters related to VAS of nausea at each recording time interval (pre-and 10, 20 and 30 min after water load) at Day 4</li> </ul> |
| Study<br>Design | <ul> <li>This is a single arm, open label pilot phase to evaluate the effect of 5-day repeated doses of exenatide (10 µg twice daily) on GMA, GE and nausea in subjects with T2DM.</li> <li>The study will comprise 3 study periods: screening/wash-out (up to 3 weeks), treatment (5 days), and post-treatment follow-up (within 7 days after the last dose of exenatide).</li> <li>The study will recruit subjects with T2DM (&gt;6 months since diagnosis) with glycated hemoglobin (HbA1c) &gt;6.5% and ≤9.0%, fasting plasma glucose (FPG) &lt;=210 mg/dL (central lab) at screening and on a current regimen of diet and exercise or a stable dose of one oral anti-diabetic medication (OAM) (maintained for &gt;= 2 months prior to screening).</li> <li>Fasting capillary blood glucose will be confirmed to be &lt;=230 mg/dL at baseline.</li> <li>Subjects receiving monotherapy with an OAM of metformin, sulfonylurea, sodium glucose co-transporter-2 (SGLT2) inhibitors, or meglitinide at screening will be washed out for 2 days for immediate release and 4 days for extended release OAM prior to baseline.</li> <li>Subject's nutritional plan will be optimized prior to baseline and</li> </ul> |

204879

| | <ul> <li>maintained during the entire study.</li> <li>All evaluations and assessments will be performed as outpatient visits. Subjects will undergo 2 EGG and 2 gastric emptying breath tests (GEBT) assessments.</li> <li>At the end of the Part A, subjects previously on an OAM will restart OAM at the discretion of the investigator after the last dose of exenatide. The half-life of exenatide (2-3 hours) should be taken into consideration.</li> <li>The total duration of a subject's participation will be approximately 5 weeks.</li> </ul> |
|---|---|
| Planned<br>Analyses | • Part A: Final Analysis: After at least 10 evaluable subjects defined as having at least one valid pre-dose EGG and one valid post –dose EGG, the final analysis for the clinical study report will be performed. At this time, the database will be frozen. The study is terminated early with a limited number of subjects enrolled in Part A. |
| Analysis<br>Populations | The analysis set will include subjects who have taken at least one dose of study medication and one valid EGG data. Data will be assessed and reviewed by the central reader before it is considered valid. |
| Hypothesis | No formal statistical hypotheses are being tested in Part A. Part A will be a pilot phase investigating the effect of repeated doses of exenatide on GMA, GE, and VAS of nausea. |
| Primary<br>Analyses | No formal statistical analyses will be performed for the exploratory endpoints for Part A. All exploratory endpoints will be assessed using descriptive statistics and graphical displays as appropriate. |

204879

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

### 2.1. Changes to the Protocol Defined Statistical Analysis Plan

The study terminated early with a limited number of subjects enrolled in Part A. Therefore, only data listings will be produced for selected data. These are limited in scope compared to the originally planned statistical analysis specified in the protocol amendment 1 [(Dated: June 23, 2016)].

### 2.2. Study Objective(s) and Endpoint(s)

#### Part A:

| Objectives | Endpoints |
|---|---|
| Exploratory Objectives | Exploratory Endpoints |
| To evaluate the effect of exenatide on GMA To assess the effect of exenatide on GE | <ul> <li>Change from baseline of EGG parameters at each recording time interval (pre-and 10, 20 and 30 min after water load) compared to baseline:</li> <li>Distribution of average power by frequency region (as % of power)</li> <li>Ratios of average power post- WLT/pre-WLT by frequency region</li> <li>Percentage (%) of time with the dominant EGG frequencies in the four frequency ranges (bradygastria, normal, tachygastria and duodenal)</li> <li>Change from baseline EGG parameters related to VAS of nausea at each recording time interval (pre-and 10, 20 and 30 min after water load) at Day 4</li> <li>Change from baseline of time to half gastric emptying (GEt½) at Day 5</li> </ul> |
| | Change from baseline of profiles of 13C excreted in breath (kPCD1) at Day 5 and at each time interval (45, 90, 120, 150, 180 and 240 min). |
| To assess the volume of water ingested during EGG | Change from baseline of volume of water ingested during EGG with water load test at Day 4. |
| To evaluate the effect of exenatide on stomach fullness, hunger, bloating and abdominal pain during EGG with water load test To evaluate safety and tolerability | Change from baseline of VAS of stomach fullness, hunger, bloating and abdominal pain during the EGG water load test at each time interval (pre-and 10, 20 and 30 min after water load) at Day 4 • Vital signs, clinical laboratory tests, AEs, |
| of exenatide | <ul><li>and GCSI-DD.</li><li>Nausea AEs presenting outside the timing of the WLT and GCSI-DD.</li></ul> |
204879

| Objectives | Endpoints |
|---|---|
| To evaluate change in gastric | At Day 4; over 30 min and at each |
| rhythm status (Data | time interval (pre-and 10, 20 and 30 min after |
| permitting) | • water load). |
| | <ul> <li>Number and % of subjects with a shift in gastric rhythm status.</li> <li>Number and % of subjects by gastric rhythm status at each time interval.</li> <li>Mean and mean change from baseline in</li> </ul> |
| | average dominant frequency |

<sup>&</sup>lt;sup>1</sup> Percent dose excreted of <sup>13</sup>C \*1000

### 2.3. Study Design

### 2.3.1. Overview of Study Design and Key Features



Due to early termination, the entirety of the study conduct was not carried out.

204879

### 2.3.2. Study Design

Part A is a single arm, open label pilot phase to evaluate the effect of 5-day repeated doses of exenatide (10  $\mu$ g twice daily) on GMA, GE and nausea in subjects with T2DM. Part A will comprise 3 study periods screening/wash-out (up to 3 weeks), treatment (5±1 days), and post-treatment follow-up (within 7 days after the last dose of exenatide).

At the time the RAP is being prepared, the study is terminated early with a limited number of subjects enrolled in Part A.

204879

#### 3. PLANNED ANALYSES

### 3.1. Interim Analyses

No interim analysis is planned for this study. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential step:

All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

### 4. ANALYSIS POPULATIONS

| Part A: | Comprise of all subjects who have taken | Pharmacodynamic |
|---|---|---|
| Pharmacodynami | at least one dose of study medication and | · |
| c | one valid EGG data Data will be assessed | |
| | and reviewed by the central reader before | |
| | it is considered valid. The central reader | |
| | will provide the valid data that will be | |
| | used for the analyses. | |
| All Subjects | All subjects with at least one dose of | Safety |
| | study medication. | |
| Enrolled | All enrolled subjects. | Enrolled |

#### NOTES:

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

### 5.1. Reporting Conventions

- All data displays will be presented according to the Integrated Data Standards Library (IDSL) reporting standards, where applicable.
- Analyses will be performed using the 9.1.3 version of the SAS System or higher (SAS is a registered trademark of the SAS Institute Inc., Cary, NC, USA).
   Programs will be imported into HARP and the final output will be produced by running drivers in HARP.
- Data collected at unplanned (i.e. unscheduled) time points will not be included
  in the summaries by visit unless otherwise stated. Unscheduled or unplanned
  readings will be presented in the listings and they will be included when
  determining worst-case flagging for post-baseline summaries.
- In all data displays, planned and actual relative times will be relative to the study drug dosing time of the relevant dosing session.

Please refer to Appendix 5: List of Data Displays which details the population to be used for each displays being generated.

204879

- Refer to IDSL standards (when applicable) for decimal place conventions. Raw data will generally be presented to the same number of decimal places as it was collected.
- All data will be reported according to the actual treatment the subject received. Any departures from the planned treatment according to the randomization schedule will be documented in the report.
- All observations that occurred prior to dosing will be considered as part of the pre-dose period. All observations that occur during dosing will be attributed to the subject's treatment.

Deviations from the analyses in the RAP will be identified in the final clinical study report.

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---------|-----------------------------------------------------|
| 9.1 | Appendix 1: Time & Events |
| 9.2 | Appendix 2: Assessment Windows |
| 9.3 | Appendix 3: Values of Potential Clinical Importance |
| 9.4 | Appendix 4: Abbreviations and Trademarks |
| 9.5 | Appendix 5: List of Data Displays |

#### 6. STUDY POPULATION ANALYSES

### 6.1. Overview of Planned Analyses

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 5: List of Data Displays.

204879

Table 2 Overview of Planned Study Population Analyses

| Display Type | Data | Data Display's Generated | |
|---|---|---|---|
| | Figure | Table | Listing |
| Subject Disposition | | | |
| Reasons for Withdrawal from Study | | Υ | Υ |
| Demography and Baseline Characteristics | | | |
| Demographics and Baseline Characteristics | | Y | Y |
| Race & Racial Combinations | | Y | Y |
| Number of subjects by Site ID | | Y | Y |
| Age Ranges | | Y | |
| Medical Condition & Concomitant Medications | | | |
| Concomitant Medication | | | Y |
| Exposure | | | |
| Exposure to Study Drug | | | Υ |

Note: additional tables, listings and figures will be provided in Appendix 5: List of Data Displays.

Following review of the data, additional analyses maybe conducted to further support the evaluation and interpretation of the data.

### 6.2. Demographic and Baseline Characteristics

Continuous variables such as age, body mass index, weight, and height will be summarized using descriptive statistics (n, mean, standard deviation, and median, minimum, maximum). Categorical variables including sex, race, ethnicity, and baseline weight category (<90 kg or  $\ge$ 90 kg) will be summarized using numbers and percentages. Continuous variables such as age, body mass index, weight, and height will be presented in a by-subject listing. Listings will be presented using the safety population, if appropriate.

#### 6.3. Exposure to Study Drug

A by-subject listing of study drug administration will also be presented. Overall study drug administration and treatment compliance will be present with the exposure to study drug listing.

#### 6.4. Medications

Any prior and concomitant medication used during the study will be recorded and coded using GSKDrug Dictionary (GSKDRUG), which will be updated whenever available throughout the life of the study.

Any medication used during the study will be recorded, which will be updated whenever available throughout the life of the study.

<sup>•</sup> Y = Yes display generated.

204879

All medications will be listed.

#### 6.5. Safety Analyses

#### 6.5.1. Overview of Planned Analyses

The safety analyses will be based on all subjects population. Table 3 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 5: List of Data Displays.

Table 3 Overview of Planned Safety Analyses

| | | Obse | erved | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| Endpoints | Sum | mary | Individ | ual | Sumi | mary | Individual | |
| | Т | F | F | L | Т | F | F | L |
| Adverse Events | Y | | | Υ | | | | |
| Clinical Laboratory | | | | Υ | | | | |
| Vital Signs | | | | Υ | | | | |
| GCSI-DD | | | | Υ | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

Following review of the data, additional analyses maybe conducted to further support the evaluation and interpretation of the data.

#### 6.5.2. Adverse Events

All AEs will be coded using MedDRA which will be updated whenever available throughout the life of the study.

All AEs will be listed in a subject data listing.

#### 6.5.3. Clinical Laboratory Evaluations

#### 6.5.3.1. Chemistry, Hematology and Urinalysis

Laboratory parameters include the following tests: hematology, chemistry and urinalysis. Established or generally acknowledged methods, normal ranges, and quality control procedures will be supplied by central lab for the study records.

Hematology parameters include red blood count, hemoglobin, hematocrit white blood cell count with differential, and platelet count. Chemistry blood urea nitrogen (BUN), potassium, aspartate aminotransferase (AST), total and direct bilirubin, creatinine, sodium, ALT, total protein, calcium, magnesium, chloride, phosphorus albumin, , gamma glutamyl transferase (GGT), estimated glomerular filtration rate (eGFR), and lipids

204879

(including total cholesterol, LDL-C, HDL C, triglycerides,). Urinalysis parameters include microalbumin and creatnine and specific gravity, pH, glucose, nitrates, leukocytes esterase, blood and ketones by dipstick and microscopic examination (if blood or protein is abnormal).

All laboratory parameters as collected will be presented in by-subject listings at every scheduled assessment time point. All listings will be done for the safety population and all laboratory data will be listed including other laboratory tests, such as TSH, and urine pregnancy test results.

Additionally, the number of subjects with laboratory values of potential clinical concern will be provided in a listing by treatment group and scheduled assessment time point for hematology and chemistry. The criteria for laboratory values of potential clinical concern are detailed in Appendix 3: Values of Potential Clinical Importance.

A listing of laboratory values of potential clinical concern will be provided for liver function tests, including ALT, AST, and total bilirubin. The criteria for liver function tests of potential clinical concern are detailed in Appendix 3: Values of Potential Clinical Importance.

#### 6.5.4. Vital Signs

The vital sign analysis will include systolic blood pressure (mmHg), diastolic blood pressure (mmHg), and heart rate (bpm).

Each vital sign parameter at every scheduled assessment time point will be presented in by-subject listings.

All listings will be produced for all subjects population.

#### 6.5.5. Gastroparesis Cardinal Symptom Index Daily Dairy (GCSI-DD)

The GCSI-DD consists of nine symptom severity items covering the following domains: nausea/vomiting; fullness/early satiety, and bloating. In addition, the GCSI-DD contains two symptom severity items upper abdominal pain and overall rating of gastroparesis symptoms. Patients rate each symptom on a 6-point scale from 0-5 with lower scores representing less symptom severity. All questions addressed in the GCSI-DD and the overall severity question will be listed in a subject data listing and by time point.

### 7. OTHER STATISTICAL ANALYSES (EXPLORATORY)

### 7.1. Overview of Planned Analyses

The study was terminated early and therefore no analysis will be performed but data listing will be generated for all exploratory endpoint as in Appendix 5.

#### 7.2. Exploratory Analyses

Listing will be provided for all endpoints.

204879

### 8. REFERENCES

None.

204879

# 9. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 9.1 | Appendix 1: Time and Events |
| Section 9.2 | Appendix 2: Assessment Windows |
| Section 9.3 | Appendix 3: Values of Potential Clinical Importance |
| Section 9.4 | Appendix 4: Abbreviations & Trade Marks |
| Section 9.5 | Appendix 5: List of Data Displays |

204879

#### 9.1. **Appendix 1 Time & Events**

#### 9.1.1. Protocol Defined Time & Events Part A

| Procedures | | ng/Wash-O<br>(0-3 Weeks | | (5 Davis) | | | Un-<br>schedule Early | | Follow Up<br>Within 7 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | -21 to<br>Day -4 | Day -3<br>to -5 | Day -113 | Day 1 | Day 2 | Day 3 | Day 4<br>±1 day <sup>(3)</sup> | Day 5<br>±1 day <sup>13</sup> | d | Withdrawal | Days . |
| Study Visit | 1 | 3 | 2 | 3 | ě | | 4 | 5 | | - 8 | 6 |
| Informed consent | X | | | | | | | | | | |
| Inclusion and exclusion criteria | X | | Χı | | | | | | | | |
| Demography, medical/disease history | X | | | | | | | | | - 3 | |
| Enrolment into Treatment Phase | | | | X | | | | | | | |
| OAM washout <sup>2</sup> | | X | | | | | | | | | |
| GEBT3 | | | X | | | | | X12 | | | |
| EGG /water load / VAS3 | 8 | | | X11 | 9 | | X12 | | | 1 | |
| ECG | X | 7 | | | | | | | | | |
| Vital Signs | X | | X | X | | | X | X | | X | X |
| Height, Weight, BMI | X | | | | | | | | | 1 | |
| Physical exam (F, Full; B, Brief) <sup>4</sup> | F | | | | | | | В | | В | |
| Concomitant medications review | X | | X | X | | | X | | X | X | X |
| AEs, SAEs, AEs of special interest review | χ5 | | χs | X | | | X | X | X | X | X |
| PAGI-SYM <sup>6</sup> | X | * | | | | | | | | 1000 | 0.00 |
| GCSI-DD | | | X | X | | 9 | X | X | | - 3 | |
| Chemistry, hematology, urinalysis, lipids <sup>7</sup> | X | | | | | | | X | | X | |
| HbAte | X | | | | | | | | | 1 | |
| FPG | X | | X | X | | | X | X | X | X | X |
| Fasting capillary glucose at clinic <sup>8</sup> | 8 | 8 | X | X | | | X | X | | - 8 | |
| Diet/Exercise/SMBG advice/reinforcement9 | X | Х | | | | | | X | X | X | X |
| Estradiol and FSH (females only: if required) | X | | | | | | | | | | 7.00 |
| Serum/Urine pregnancy test (FRP only) | S | | U | | | | | U | | U | U |
| TSH, Amylase and lipase | X | | | | | | | | | | |
| Genetics sample <sup>10</sup> | | | | X | | | | | | | Ti di di |
| RAMOS registration | | | | X | | | | | | X | X |

| Procedures | | Screening/Wash-Out Period<br>(0-3 Weeks) | | | | | | | Follow Up |
|---|---|---|---|---|---|---|---|---|---|
| -21 to Day -3<br>Day 4 to -5 Day -1 <sup>13</sup> | Day 1 | Day 2 | Day 3 | Day 4<br>±1 day <sup>(3)</sup> | Day 5<br>±1 day <sup>13</sup> | schedule<br>d | Early<br>Withdrawal | Within 7<br>Days | |
| Study Visit | 1 | | 2 | 3 | | | 4 | 5 | 6 |
| Exenatide dosing | | | | Х11 | X | X | X12 | X12 | 1000 |
| Study medication compliance | | 83 | 0 | Y | | | Y | Y | |

Note: section noted in time and event table referring to the protocol.

Before baseline assessment (Day -1), the investigator must review all inclusion and exclusion criteria to confirm subject's eligibility. If a subject no longer meets all of the eligibility criteria, do not administer the study treatment and contact the Medical Monitor to discuss how to proceed (e.g., to determine if repeat testing is warranted). For subjects taking OAM at screening only. At a minimum, two day washout for immediate release and at minimum 4 day washout for extended release OAMs. See footnote 13. For information on restarting OAM refer to Section 6.9.

A small meal will be provided 2 hrs prior to the EGG procedure (Section 7.3.1). A meal will also be provided post-procedure for both the EGG and GEBT. Details of full and brief physical examinations are provided in Section 7.4.3.

SAEs related to study participation only.

The GCSI-DD guestionswise will be computed after the standard AE.

The GCSI-DD questionnaire will be completed after the standard AE questions have been answered.
 The GCSI-DD questionnaire will be completed after the standard AE questions have been answered.
 Clinical chemistry, hematology, urinalysis and lipid assessments are described in Section 7.4.6. Lipids will be assessed at screening only.
 Fasting capillary glucose will be measured prior to administration of exenatide. On GEBT (Day 5) or EGG (Day 1 and Day 4) assessment days, fasting capillary glucose will be measured prior to the GEBT or EGG procedure. 9. Subjects will be provided with diet and exercise guidance (see Section 7.4.9), and instructed on self monitoring blood glucose at screening (See Section 7.4.9). Subject will be

instructed to bring in their glucometers at each visit for review. Diet/exercise/SMBG reinforced at subsequent visits.

10. Informed consent for optional genetic research should be obtained before collecting a sample.

Informed consent for optional genetic research should be obtained before coinciding a sample.
 On the morning of Day 1, subjects will receive instructions and training on exenatiole self administration and will be monitored by medical staff at the clinic during administration of the first dose. The first dose of exenatide will be administered after the baseline EGG procedure and before the post-procedure meal.
 On Day 4 and 5, the morning dose of exenatide will be administered at clinic 1 hr (±15 min) before the EGG or GEBT procedure.
 Every effort should be made to schedule the procedures on the nominal visit day identified. However, in order to meet scheduling needs, subjects taking OAM can schedule Day-1 up to 3 days prior to Day 1 and the OAM stopped at least the day before the GEBT. For subjects treated with diet and exercise alone Day-1 can occur within 7 days prior to Day 1. The EGG and GEBT should not be scheduled on the same day

204879

### 9.2. Appendix 2 Assessment Windows

### 9.2.1. Definitions of Study Day

When study day is used for display or in comparisons the following algorithm will be used:

- Study day = date of assessment date of first dose + 1, if day of assessment >= first dose date
- Study day = date of assessment date of first dose, if day of assessment < first dose date

Note that the date of first dose is Day 1 and the day before the date of first dose is Day -1 (there is no Day 0).

204879

# 9.3. Appendix 3 Values of Potential Clinical Importance

# 9.3.1. Laboratory

| | Hematology | | |
|---|---|---|---|
| Laboratory<br>Test | Units | Change from Baseline of<br>Potential Clinical Concern | Potential Clinical Concern<br>Value |
| Basophils | GI/L | None | None |
| Eosinophils | GI/L | None | None |
| Hematocrit | 1 | >0.1 decrease | >0.05 below LLN<br>>0.04 above ULN |
| Hemoglobin | g/L | >25 g/L decrease | >20 g/L below LLN<br>>10 g/L above ULN |
| Lymphocytes | GI/L | None | <0.5 x LLN |
| Monocytes | GI/L | None | None |
| Neutrophils | GI/L | None | <1 GI/L |
| Neutrophil<br>Bands | GI/L | None | None |
| Platelets | GI/L | None | <80 GI/L<br>>500 GI/L |
| Red Blood Cell<br>Count | TI/L | None | None |
| Segmented<br>Neutrophils | GI/L | None | <0.5 x LLN |
| White Blood Cell<br>Count | GI/L | None | >1 GI/L below LLN<br>>5 GI/L above ULN |

| | Chemistry | | |
|---|---|---|---|
| Laboratory<br>Test | Units | Change from Baseline of<br>Potential Clinical Concern | Potential Clinical Concern<br>Value |
| Albumin | g/L | None | >5 g/L above ULN or below LLN |
| Alkaline<br>Phosphatase | U/L | None | >3 x ULN |
| ALT | U/L | None | >3 x ULN |
| AST | U/L | None | >3 x ULN |
| Bicarbonate<br>(Carbon Dioxide<br>Content) | mmol/L | None | <16 mmol/L<br>> 40 mmol/L |
| Blood Urea<br>Nitrogen | mmol/L | None | >2 x ULN |
| Calcitonin | pmol/L | None | >100 |
| Calcium | mmol/L | None | <1.8 mmol/L<br>>3.0 mmol/L |

204879

| | Chemistry | | |
|---|---|---|---|
| Laboratory<br>Test | Units | Change from Baseline of<br>Potential Clinical Concern | Potential Clinical Concern<br>Value |
| Chloride | mmol/L | None | None |
| Creatinine | umol/L | None | >159 umol/L |
| Direct Bilirubin | umol/L | None | >1.35 x ULN |
| Gamma<br>Glutamyl<br>Transferase | U/L | None | >3 x ULN |
| Glucose<br>(fasting) | mmol/L | None | <3 mmol/L<br>>22 mmol/L |
| Magnesium | mmol/L | None | <1 mmol/L<br>>4 mmol/L |
| Phosphorus | mmol/L | None | >0.323 mmol/L above ULN or below LLN |
| Potassium | mmol/L | None | >0.5 mmol/L below LLN<br>>1.0 mmol/L above ULN |
| Sodium | mmol/L | None | >5 mmol/L above ULN or below LLN |
| Total Bilirubin | umol/L | None | >1.5 x ULN |
| Total Protein | g/L | None | >15 g/L above ULN or below LLN |
| Uric acid | umol/L | None | >654 umol/L |
| Free Fatty Acids | mmol/L | None | None |
| HDL Cholesterol | mmol/L | None | None |
| LDL Cholesterol | mmol/L | None | None |
| Triglycerides | mmol/L | None | > 9.04 mmol/L |
| Total<br>Cholesterol | mmol/L | None | None |

204879

| I shouston. Test | Detection Official Company Value |
|------------------|-----------------------------------------|
| Laboratory Test | Potential Clinical Concern Value |
| ALT | ≥2 x ULN |
| | ≥ 3 x ULN |
| | ≥ 5 x ULN |
| | ≥8 x ULN |
| | ≥ 10 x ULN |
| | ≥ 3 x ULN and Total Bilirubin ≥ 2 x ULN |
| AST | ≥ 2 x ULN |
| | ≥ 3 x ULN |
| | ≥ 5 x ULN |
| | ≥8 x ULN |
| | ≥ 10 x ULN |
| | ≥ 3 x ULN and Total Bilirubin ≥ 2 x ULN |
| Total Bilirubin | ≥ 1.5 x ULN |
| | ≥ 2 x ULN |
| | ≥ 3 x ULN |
| | ≥ 5 x ULN |
| | ≥8 x ULN |
| | ≥ 10 x ULN |

204879

# 9.4. Appendix 4 – Abbreviations & Trade Marks

### **Abbreviations**

| ADA | American Diabetes Association |
|-------------|--------------------------------------------------------|
| AE | adverse event |
| ALT (SGPT) | alanine aminotransferase (serum glutamic pyruvic |
| TIET (SGIT) | transaminase) |
| AST (SGOT) | aspartate aminotransferase (serum glutamic oxaloacetic |
| 1101 (5001) | transaminase) |
| BMI | body mass index |
| BUN | blood urea nitrogen |
| CI | confidence interval |
| CONSORT | Consolidated Standards of Reporting Trials |
| CPK | creatine phosphokinase |
| CV | cardiovascular |
| DCC | dual chamber cartridge |
| DNA | deoxyribonucleic acid |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| eGFR | estimated glomerular filtration rate |
| EGG | electrogastrogram |
| ELISA | enzyme-linked immunosorbent assay |
| EMA | European Medicines Agency |
| FDA | US Food and Drug Administration |
| FFA | free fatty acids |
| FPG | fasting plasma glucose |
| FRP | females of reproductive potential |
| FSH | follicle stimulating hormone |
| GCP | Good Clinical Practice |
| GCSP | Global Clinical Safety and Pharmacovigilance |
| GGT | gamma glutamyl transferase |
| GI | gastrointestinal |
| GLP-1 | glucagon-like peptide-1 |
| GSK | GlaxoSmithKline |
| НА | human albumin |
| HbA1c | glycated hemoglobin |
| HBcAb | hepatitis B core antibody |
| HBsAg | hepatitis B surface antigen |
| HIV | human immunodeficiency virus |
| hCG | human chorionic gonadotrophin |
| HDL-c | high density lipoproteins |
| HRP | horseradish peroxidase |
| HRT | hormone replacement therapy |

204879

| IB | Investigator's Brochure |
|---|---|
| ICH | International Conference on Harmonization |
| IEC | Independent Ethics Committee |
| INR | international normal range |
| IP IP | investigational product |
| IRB | Institutional Review Board |
| ISRs | injection site reactions |
| ITT | 3 |
| IVRS | intent-to-treat Interactive Voice Response System |
| LDH | lactate dehydrogenase |
| LDL-c | low density lipoproteins; |
| LMCF | last mean carried forward |
| K <sub>2</sub> EDTA | di-potassium ethylenediaminetetraacetic acid |
| MACE | major adverse cardiovascular event |
| MCH | mean corpuscular hemoglobin |
| MCV | mean corpuscular volume Modification of Diet in Renal Disease |
| MDRD | |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MEN-2 | multiple endocrine neoplasia type 2 |
| MI | myocardial infarction |
| MSDS | Material Safety Data Sheet |
| MTC | medullary thyroid cancer |
| OC RDC | Oracle Clinical Remote Data Capture |
| PAC | Pancreatitis Adjudication Committee |
| PD | pharmacodynamics |
| PK | pharmacokinetics |
| PP | per protocol |
| PTS-DPMK | Platform Technologies and Science-Drug Metabolism and |
| | Pharmacokinetics |
| RAP | Reporting Analysis Plan |
| RBC | red blood cell |
| RNA | ribonucleic acid |
| s.c. | subcutaneous |
| SAC | Statistical Analysis Complete |
| SAE | serious adverse event |
| SmPC | Summary of Product Characteristics |
| SRM | Study Reference Manual |
| SU | sulfonylureas |
| T2DM | type 2 diabetes mellitus |
| TSH | thyroid stimulating hormone |
| ULN | upper limit of normal range |
| WBC | white blood cell |
| WCBP | women of child bearing potential |

204879

### **Trademark Information**

Trademarks of the GlaxoSmithKline group of companies

NONE

Trademarks not owned by the GlaxoSmithKline group of companies

MedDRA

204879

# 9.5. Appendix 5 List of Data Displays

# 9.5.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Listings | Tables |
|-----------------------|----------|------------|
| Study Population | 1 to 5 | 1.1 to 1.5 |
| Safety | 6 to 14 | 1.6 to 1.7 |
| Exploratory Endpoints | 15 | |

### 9.5.2. Study Population Tables

| Stud | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No | Popula<br>tion | IDSL /<br>TST ID /<br>Exampl<br>e Shell | Title | Programming Notes | Delivera<br>ble<br>[Priority] |
| [Dis | position] | | | | |
| 1.1. | All<br>Subject<br>s | ES1/ES<br>1A | Summary of Subjects Disposition for the Subject Conclusion Record | | |
| [Den | nographics | and Base | ine Characteristics] | | |
| 1.2. | All<br>Subject<br>s | DM1 | Summary of Demographic Characteristics | | |
| 1.3. | All<br>Subject<br>s | DM5 | Summary of Race & Racial Combinations | | |
| 1.4. | Enrolle<br>d | NS1 | Summary of Number of Subjects by Country and Site ID | | |
| 1.5. | Enrolle<br>d | DM11 | Summary of Age Ranges | | |
| Safe | ty Tables | | | | |
| 1.6. | All<br>Subject<br>s | AE15 | Summary of Common (>=2%) Non-<br>serious AEs by System Organ Class<br>and Preferred Term | | |
| 1.7. | All<br>Subject<br>s | AE16 | Summary of Serious AEs by System<br>Organ Class and Preferred Term | | |

204879

# 9.5.3. Listings

| Listi | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 1. | All Subjects | | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | |
| 2. | All Subjects | | Listing of Reasons for Withdrawal from Study | | |
| 3. | All Subjects | | Listing of Demographics and Baseline Characteristics | | |
| 4. | All Subjects | | Listing of Race | | |
| 5. | All Subjects | | Listing of Subjects by Site ID | | |
| 6. | All Subjects | | Listing of Concomitant<br>Medication by Generic Term | | |
| 7. | All Subjects | | Listing of All Adverse Events | | |
| 8. | All Subjects | | Listing of Hematology<br>Laboratory Data | | |
| 9. | All Subjects | | Listing of Chemistry<br>Laboratory Data | | |
| 10. | All Subjects | | Listing of Urinalysis Laboratory Data | | |
| 11. | All Subjects | | Listing of Laboratory Data for<br>Subjects with Any Value of<br>Potential Clinical Concern | | |
| 12. | All Subjects | | Listing of Liver Functions with<br>Any Value of Potential Clinical<br>Concern | | |
| 13. | All Subjects | | Listing of Vital Signs | | |
| 14. | All Subjects | | Listing of GCSI-DD | | |
| 15. | Pharmacodynamic | | Listing of all EGG endpoints. | | |